CLINICAL TRIAL: NCT02960997
Title: A Prospective, Double-Blind, Cross-Over, Pilot Study to Assess Safety and Efficacy of Topical Sirolimus 2% in the Treatment of Plantar Blistering in Patients With Epidermolysis Bullous Simplex (EBS)
Brief Title: Using Topical Sirolimus 2% for Patients With Epidermolysis Bullous Simplex (EBS) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Joyce Teng, Director of Pediatric Dermatology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 35498
Record Dates: First submitted 2016-06-15; First posted 2016-11-10 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Epidermolysis Bullosa Simplex; Epidermolysis Bullosa Simplex Kobner; Weber-Cockayne Syndrome
Keywords: epidermolysis bullosa simplex
MeSH Terms: conditions — Epidermolysis Bullosa Simplex | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus, then Placebo (Experimental): Participants will receive Sirolimus, 2% topical ointment for 12 weeks followed by placebo to match sirolimus for 12 weeks.
  Interventions: Drug: Sirolimus, 2%; Drug: Vehicle
- Placebo, then Sirolimus (Placebo Comparator): Participants will receive placebo to match sirolimus for 12 weeks followed by Sirolimus, 2% topical ointment for 12 weeks.
  Interventions: Drug: Sirolimus, 2%; Drug: Vehicle

INTERVENTIONS:
Drug: Sirolimus, 2%
Drug: Vehicle
  Other Names: Placebo

SUMMARY:
Epidermolysis bullosa (EB) simplex is a rare orphan disease caused by a mutation in DNA leading to abnormal dominant keratins in the skin. Patients with EB simplex develop lifelong painful thick soles on their feet, and current standard of care is supportive. This pilot study will target the dominant mutant keratin proteins in the skin to ameliorate the severity of EB simplex. The purpose is to improve the function of EB simplex feet with an application of topical sirolimus, 2%. The investigators plan on inhibiting the mTOR pathway to down regulate the translation of defective keratin proteins and work through anti proliferative pathways.

DETAILED DESCRIPTION:
The proposed 40 week pilot study being conducted is a prospective, double-blind, randomized, placebo-controlled crossover study. Participants will be assigned to treat both feet with either topical sirolimus, 2% cream daily or placebo (vehicle-control) for 12 weeks, followed by a 4 week washout period, then re-treatment to both feet will occur by the cross-over intervention.

These studies will exploit the naturally occurring transcriptional regulation of keratin sequences, the known gene aberration causing EB simplex, and assess the potential for mTOR pathway inhibition in treatment of the patient's plantar lesions. The objective of this study is to assess (1) the safety of topical rapamycin for plantar lesions for the treatment of EB simplex, and 2) test if topical rapamycin to improves the clinical severity of lesional skin, including pain and itch, in subjects with EB simplex at the end of treatment versus baseline and compared to an intrasubject placebo treated control. Wound size measurement, quality of life evaluation will be assessed using epidermolysis bullosa (QOLEB), and EB disease activity and Scarring Index (EBDASI). With the results of this pilot study, physicians would be able to transition from supportive care (the current state of the art for EB simplex) to targeted molecular therapeutics, leading to improved mobility and quality of life for patients with EB simplex.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* Be capable of understanding the purpose and risks of the study and sign a written Informed Consent Form (ICF); Legally authorized representative of subjects willing and able to give consent for children 4-18 yo.
* Be male or female with a diagnosis of EBS
* Minimum EBDASI feet activity score of 2/10
* Age - 4 years or older
* Ability to complete 12 study visits within a 40-week period, each for approximately 30-60 minutes.
* Anticipated life expectancy ≥52 weeks.
* Males and females of childbearing potential should be using an effective means of contraception.
* Laboratory values within the range of normal for the participating institution unless the PI feels they are not clinically relevant
* Be able to comply with all study requirements

Exclusion Criteria:

* Allergy to sirolimus or components of the vehicle ointment
* Pregnancy, breast feeding
* Prior history of liver disease
* Serious known concurrent medical illness or infection, which could potentially present a safety risk and/or prevent compliance with the requirements of the treatment program.
* Known immunodeficiency virus or syndrome including those with:

  * Acquired Immunodeficiency Syndrome (AIDS)
  * Human Immunodeficiency Virus (HIV)
  * Hepatitis B
* Prior history of grafting surgeries or other surgeries in the dermatologic treatment area
* History of significant condition in the dermatologic treatment area such as trauma, which could impair evaluation for the treatment of EBS or non-healing chronic wound.
* Use of other investigational drugs within 30 days of the screening visit and/or has not recovered from any side effects of prior investigational drugs or procedure in the affected area (e.g., a biopsy).
* Use of acitretin within the last 1 month
* Use of Roaccutane within last 3 months
* Botox injections to the feet within the last 6 months.
* Participant is planning extra physical activities within the next 3 months.
* Amputated foot

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12-14 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce M Teng, MD, PhD, Study Chair — Stanford School of Medicine
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fine JD, Bruckner-Tuderman L, Eady RA, Bauer EA, Bauer JW, Has C, Heagerty A, Hintner H, Hovnanian A, Jonkman MF, Leigh I, Marinkovich MP, Martinez AE, McGrath JA, Mellerio JE, Moss C, Murrell DF, Shimizu H, Uitto J, Woodley D, Zambruno G. Inherited epidermolysis bullosa: updated recommendations on diagnosis and classification. J Am Acad Dermatol. 2014 Jun;70(6):1103-26. doi: 10.1016/j.jaad.2014.01.903. Epub 2014 Mar 29. PMID 24690439
- [Background] Fine JD, Johnson LB, Weiner M, Suchindran C. Assessment of mobility, activities and pain in different subtypes of epidermolysis bullosa. Clin Exp Dermatol. 2004 Mar;29(2):122-7. doi: 10.1111/j.1365-2230.2004.01428.x. PMID 14987264
- [Background] Lane EB, McLean WH. Keratins and skin disorders. J Pathol. 2004 Nov;204(4):355-66. doi: 10.1002/path.1643. PMID 15495218
- [Background] Castedo M, Ferri KF, Kroemer G. Mammalian target of rapamycin (mTOR): pro- and anti-apoptotic. Cell Death Differ. 2002 Feb;9(2):99-100. doi: 10.1038/sj.cdd.4400978. No abstract available. PMID 11840159
- [Background] Guba M, von Breitenbuch P, Steinbauer M, Koehl G, Flegel S, Hornung M, Bruns CJ, Zuelke C, Farkas S, Anthuber M, Jauch KW, Geissler EK. Rapamycin inhibits primary and metastatic tumor growth by antiangiogenesis: involvement of vascular endothelial growth factor. Nat Med. 2002 Feb;8(2):128-35. doi: 10.1038/nm0202-128. PMID 11821896
- [Background] Fogel AL, Hill S, Teng JM. Advances in the therapeutic use of mammalian target of rapamycin (mTOR) inhibitors in dermatology. J Am Acad Dermatol. 2015 May;72(5):879-89. doi: 10.1016/j.jaad.2015.01.014. Epub 2015 Mar 11. PMID 25769191
- [Background] Raught B, Gingras AC, Sonenberg N. The target of rapamycin (TOR) proteins. Proc Natl Acad Sci U S A. 2001 Jun 19;98(13):7037-44. doi: 10.1073/pnas.121145898. PMID 11416184
- [Background] Hickerson RP, Leake D, Pho LN, Leachman SA, Kaspar RL. Rapamycin selectively inhibits expression of an inducible keratin (K6a) in human keratinocytes and improves symptoms in pachyonychia congenita patients. J Dermatol Sci. 2009 Nov;56(2):82-8. doi: 10.1016/j.jdermsci.2009.07.008. Epub 2009 Aug 21. PMID 19699613
- [Background] Riskowski JL, Hagedorn TJ, Hannan MT. Measures of foot function, foot health, and foot pain: American Academy of Orthopedic Surgeons Lower Limb Outcomes Assessment: Foot and Ankle Module (AAOS-FAM), Bristol Foot Score (BFS), Revised Foot Function Index (FFI-R), Foot Health Status Questionnaire (FHSQ), Manchester Foot Pain and Disability Index (MFPDI), Podiatric Health Questionnaire (PHQ), and Rowan Foot Pain Assessment (ROFPAQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S229-39. doi: 10.1002/acr.20554. No abstract available. PMID 22588747
- [Background] Loh CC, Kim J, Su JC, Daniel BS, Venugopal SS, Rhodes LM, Intong LR, Law MG, Murrell DF. Development, reliability, and validity of a novel Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI). J Am Acad Dermatol. 2014 Jan;70(1):89-97.e1-13. doi: 10.1016/j.jaad.2013.09.041. PMID 24355263
- [Background] Venugopal SS, Yan W, Frew JW, Cohn HI, Rhodes LM, Tran K, Melbourne W, Nelson JA, Sturm M, Fogarty J, Marinkovich MP, Igawa S, Ishida-Yamamoto A, Murrell DF. A phase II randomized vehicle-controlled trial of intradermal allogeneic fibroblasts for recessive dystrophic epidermolysis bullosa. J Am Acad Dermatol. 2013 Dec;69(6):898-908.e7. doi: 10.1016/j.jaad.2013.08.014. Epub 2013 Sep 24. PMID 24075228
- [Background] Frew JW, Martin LK, Nijsten T, Murrell DF. Quality of life evaluation in epidermolysis bullosa (EB) through the development of the QOLEB questionnaire: an EB-specific quality of life instrument. Br J Dermatol. 2009 Dec;161(6):1323-30. doi: 10.1111/j.1365-2133.2009.09347.x. Epub 2009 Jun 11. PMID 19681875
- [Background] Elman S, Hynan LS, Gabriel V, Mayo MJ. The 5-D itch scale: a new measure of pruritus. Br J Dermatol. 2010 Mar;162(3):587-93. doi: 10.1111/j.1365-2133.2009.09586.x. Epub 2009 Dec 1. PMID 19995367
- [Background] Storm FA, Heller BW, Mazza C. Step detection and activity recognition accuracy of seven physical activity monitors. PLoS One. 2015 Mar 19;10(3):e0118723. doi: 10.1371/journal.pone.0118723. eCollection 2015. PMID 25789630

RESULTS

PARTICIPANT FLOW:
Period: First Intervention, 12 Weeks
Arm/Group | Sirolimus, Then Placebo | Placebo, Then Sirolimus
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Washout Period, 4 Weeks
Arm/Group | Sirolimus, Then Placebo | Placebo, Then Sirolimus
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Second Treatment, 12 Weeks
Arm/Group | Sirolimus, Then Placebo | Placebo, Then Sirolimus
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Follow-up Period, 4 Weeks
Arm/Group | Sirolimus, Then Placebo | Placebo, Then Sirolimus
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus, Then Placebo | Placebo, Then Sirolimus | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 3
  Hispanic | 1 | 3 | 4
  Black | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8
Foot Health Status Questionnaire, Foot Function [Mean (Standard Deviation); unit: score on a scale] — Low Score (0) means severely limited in performing a broad range of physical activities. High Score (100) means can perform all desired physical activities. Data are reported according to randomization group.
  score on a scale | 51.6 (11.16) | 51.6 (20.90) | 51.6 (16.76)
Foot Health Status Questionnaire, Physical Activity [Mean (Standard Deviation); unit: score on a scale] — Low Score (0) means severely limited in performing a broad range of physical activities. High Score (100) means can perform all desired physical activities. Data are reported according to randomization group.
  score on a scale | 63.9 (25.00) | 54.2 (22.35) | 59.0 (24.21)
Child Dermatological Quality of Life Questionnaire [Mean (Standard Deviation); unit: score on a scale] — Quality of Life-Epidermolysis Bullosa (QOLEB) scores range from 0 to 51; higher scores indicate greater impact of EB on quality of life. Data are reported according to randomization group.
  score on a scale | 18.0 (10.17) | 17.3 (4.60) | 17.6 (7.90)
Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) Disease Severity Scale [Mean (Standard Deviation); unit: score on a scale] — Scores range from 0 (absent of EB) to 10 (entire area involved). Data are reported according to randomization group.
  score on a scale | 2.8 (0.43) | 3.5 (0.87) | 3.1 (0.78)
5-D Pruritus Score [Mean (Standard Deviation); unit: score on a scale] — Total score ranges from 5 (least affected) to 25 (most affected). Data are reported according to randomization group.
  score on a scale | 15.0 (1.87) | 11.0 (2.35) | 13.0 (2.92)

OUTCOME MEASURES:

1. Primary Outcome: Foot Health Status Questionnaire, Foot Function Domain Score
Description: Foot function was assessed utilizing the validated Foot Health Status Questionnaire (FHSQ). Low Score (0) means severely limited in performing a broad range of physical activities. High Score (100) means can perform all desired physical activities. Data are reported per intervention.
Time Frame: Week 0 and week 12 of the respective treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sirolimus: Sirolimus, 2% topical ointment for 12 weeks
- Placebo: Placebo to match sirolimus for 12 weeks
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale
  Week 0 | 61.7 (26.48) | 49.3 (20.83)
  Week 12 | 60.2 (23.37) | 56.3 (24.09)

2. Primary Outcome: Foot Health Status Questionnaire, Physical Activity Domain Score
Description: Physical Activity was assessed utilizing the validated Foot Health Status Questionnaire (FHSQ). Low Score (0) means severely limited in performing a broad range of physical activities. High Score (100) means can perform all desired physical activities. Data are reported per intervention.
Time Frame: Week 0 and week 12 of the respective treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale
  Week 0 | 69.4 (24.37) | 54.2 (21.65)
  Week 12 | 70.8 (20.37) | 61.8 (24.91)

3. Primary Outcome: Trough Concentration of Sirolimus
Description: Trough measurements were taken prior to topical sirolimus administration at the week 12 study visit.
Time Frame: Week 12
Population: Trough concentration of sirolimus was collected during Sirolimus treatment only, so the Placebo group is not presented in this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sirolimus
Number analyzed (Participants) | 8
ng/mL | NA (NA) — All measurements were below the lower limit of quantitation (<2 ng/mL).

4. Secondary Outcome: Average Steps Per Day Assessed by FitBit® / Pedometer
Description: Average number of steps walked per day from baseline to the end of each treatment.
Time Frame: 12 weeks
Population: One participant had no Fitbit data during placebo treatment and is excluded from the analysis. Three participants lost their Fitbit devices for week 12 reporting during sirolimus treatment; their data through week 8 are included in the analysis.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 8 | 7
steps | 6624 (1847) | 7130 (3025)

5. Secondary Outcome: Child Dermatological Quality of Life Questionnaire Score
Description: Quality of Life-Epidermolysis Bullosa (QOLEB) Questionnaire specifically designed for people with EB. The QOLEB can be used to identify everyday life occurrences negatively affected by EB. It assesses change in quality of life over time, an important measure when assessing the success of new treatments for EB. Scores from 0 to 51, with higher scores indicate greater impact of EB on quality of life. Data are reported per intervention.
Time Frame: Week 0 and week 12 of the respective treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale
  Week 0 | 14.1 (9.37) | 6.6 (8.79)
  Week 12 | 14.5 (10.14) | 13.3 (9.32)

6. Secondary Outcome: Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) Disease Severity Scale Score
Description: The EBDASI is a validated scoring system that objectively quantifies the severity of EB affecting the entire body. It has been designed to evaluate the response to new therapies for the treatment of EB. Scores range from 0 (absent of EB) to 10 (entire area involved). Data are reported per intervention.
Time Frame: Week 0 and week 12 of the respective treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale
  Week 0 | 2.6 (1.32) | 3.5 (1.22)
  Week 12 | 2.9 (1.54) | 2.5 (1.41)

7. Secondary Outcome: 5-D Pruritus Scale Score
Description: The 5-D Pruritus Scale is a 1-page, 5-question tool used in clinical trials to assess 5 dimensions of background itch: degree, duration, direction, disability, and distribution. Each question corresponds to 1 of the 5 dimensions of itch; participants were to rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected. After the summation of individual score, the total score ranges from 5 (least affected) to 25 (most affected). Data are reported per intervention.
Time Frame: Week 0 and week 12 of the respective treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale
  Week 0 | 12.8 (3.03) | 11.5 (1.87)
  Week 12 | 12.5 (3.46) | 11.8 (3.80)

8. Secondary Outcome: Plantar Defect Size Using 3D Photography
Description: Plantar defect size measurements using 3D photography (% change in total defect area).
Time Frame: Baseline, week 12
Population: Data were not collected for this outcome measure.
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Foot Plantar Pressure Measurements
Description: Foot plantar pressure measurements before and after treatment using the Podotech Elftman Foot Scanner.
Time Frame: Baseline, week 12
Population: Data were not collected for this outcome measure.
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in mTOR Pathway Inhibition
Description: Molecular biology study of skin biopsies assayed for mTOR pathway inhibition (e.g. determination of phosphoprotein inhibition included ribosomal protein S6, S6 kinase and/or eIF-4E binding protein).
Time Frame: Baseline, week 12
Population: Data were not collected for this outcome measure
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Sirolimus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=8) | Placebo (N=8)
Allergic Reaction to antiobiotic (sulfamethoxole) (Immune system disorders) | 0 | 1
Burning sensation on feet (Skin and subcutaneous tissue disorders) | 1 | 0
Common cold (Infections and infestations) | 0 | 3
Cough (General disorders) | 0 | 2
Ear infection (Infections and infestations) | 2 | 0 — 1 event occurred during the follow-up period
Feet pain (General disorders) | 1 | 1
Food poisioning (Injury, poisoning and procedural complications) | 0 | 1
High fever (Infections and infestations) | 1 | 0
Increased foot pain (General disorders) | 0 | 2
Leg infected lesion (Infections and infestations) | 1 | 0
Loose stool (Gastrointestinal disorders) | 0 | 1
Painful urination (Renal and urinary disorders) | 1 | 0
Right and left leg abrasion (Injury, poisoning and procedural complications) | 0 | 1
Right footstaph infection (Infections and infestations) | 0 | 1
Right thigh abrasion (Injury, poisoning and procedural complications) | 0 | 1
Seasonal allergies (Immune system disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upset stomach (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT02960997/Prot_SAP_000.pdf